CLINICAL TRIAL: NCT00283023
Title: Phase 1: Oligodendrocyte Progenitor Cell Culture From Human Brain
Brief Title: Oligodendrocyte Progenitor Cell Culture From Human Brain
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Responsible Party: Assistant Professor Subsai Kongsaengdao, Rajavithi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RH-CMR-003; RVH-CMR-003 grant
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Demyelinating Diseases
Keywords: All selective craniotomy
MeSH Terms: conditions — Demyelinating Diseases | interventions — Craniotomy

STUDY DESIGN:
Intervention Model Description: Cell culture
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Progenitor cells from the patinets with Craniotomy with V-P Shunt or ventriculostomy will be collected and cultured.
  Interventions: Procedure: Oligodendrocyte progenitor cell culture/craniotomy

INTERVENTIONS:
Procedure: Oligodendrocyte progenitor cell culture/craniotomy — Oligodendrocyte progenitor cell culture protocol of Rajavithi Hospital will be apply
  Other Names: Rajavithi Oligodendrocyte progenitor cell culture protocol

SUMMARY:
Recent developments in the understanding of stem- and progenitor cell differentiation raises hopes that brain damage in chronic neurological diseases may become repaired by systemic or focal transplantation of such cells. Clinical trials of stem- or progenitor cell transplantation in multiple sclerosis are currently premature. The researchers developed a protocol for human oligodendrocyte progenitor cell culture from human brain for the treatment of demyelinating disease.

DETAILED DESCRIPTION:
Oligodendrocyte progenitor cell line were cultures and will be transplanted into the patient with Multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 20-65 years of age
* Informed consent
* Has elective craniotomy surgery

Exclusion Criteria:

* HIV, hepatitis, and other central nervous system (CNS) infections
* Dementia, Alzheimer disease, and neurodegenerative disease

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-12 (Actual); Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Number of oligodendrocyte progenitor cell differentiation | one month

CONTACTS AND LOCATIONS:
Overall Officials: Subsai Kongsaengdao, M.D., Principal Investigator — Division of Neurology, Department of Medicine, Rajavithi Hospital : Thailand
Locations (1):
- Assistant Professor Subsai Kongsaengdao, Bangkok, Thailand